CLINICAL TRIAL: NCT02262273
Title: Real-World Treatment Patterns, BRCA Testing Practices, Outcomes, and Health Care Utilization in Platinum-Sensitive Recurrent Serous Ovarian Cancer: A Multi-Country Retrospective Study
Brief Title: OSCA - Olaparib Standard of CAre Study
Acronym: OSCA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: RTI Health Solutions (Other); A+A Healthcare Marketing Research (Industry); Freelance CRA (FCRA) (Unknown)
Responsible Party: Sponsor
Other Study IDs: D0816R00004
Record Dates: First submitted 2014-10-06; First posted 2014-10-13 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Platinum-sensitive Recurrent Serous Ovarian Cancer
Keywords: women; platinum sensitive; recurrent; serous; ovarian cancer; BRCA; PARP; Olaparib
MeSH Terms: conditions — Recurrence; Ovarian Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Serous ovarian cancer:: Women with platinum-sensitive recurrent serous ovarian cancer
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — Colleciton of data from medical records only

SUMMARY:
This study will be carried out as a retrospective, non-interventional observational review of medical records for patients in multiple countries with platinum-sensitive recurrent serous ovarian cancer. The objectives are to describe in a real-world population, treatment patterns, BRCA mutation testing and results, overall survival, health care utilization and also to estimate rates of selected treatment- and/or disease-related side effects

ELIGIBILITY:
Inclusion Criteria:

1. First determined to have platinum-sensitive recurrent serous ovarian cancer between January 1, 2009, and December 31, 2013 (study entry period), as defined by no evidence of disease progression for at least 6 months after completion of a first-line platinum-based chemotherapy regimen; the first date of platinum-sensitive recurrence between January 1, 2009 and December 31, 2013 will define the study index date.
2. At least 18 years of age on the index date.
3. Fully documented medical history related to the patient's ovarian cancer treatment beginning with initial diagnosis of serous ovarian cancer.
4. Patients can be either alive or deceased at the time of medical record abstraction.

Exclusion Criteria:

1. Ever taken an investigational product as part of an interventional clinical trial for ovarian cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: platinum-sensitive recurrent serous ovarian cancer patients
Sampling Method: Probability Sample
Enrollment: 2123 (Actual)
Dates: Start 2014-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Best response to therapy and date of response for each subsequent therapy line post-index | Data will be collected retrospectively from medical records
  Response categories: complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD) Criteria on which physicians determined therapy response also will be captured (e.g., symptoms, radiological and/or other imaging findings, CA-125 levels, physical exam, or other criteria).

SECONDARY OUTCOMES:
Progression-free survival, by therapy line | Data will be collected retrospectively from medical records
  Defined as time from initiation of the therapy line (including the required first-line platinum-based chemotherapy) until the earliest of progression, death, or end of follow-up (for censored observations) Criteria on which physicians determined progression also will be captured (e.g., symptoms, radiological and/or other imaging findings, CA-125 levels, physical exam, or other criteria)
Overall survival, calculated from various time points | Data will be collected retrospectively from medical records
  From first diagnosis of ovarian cancer until death or end of follow-up, whichever is earliest From initiation of the required first-line platinum-based chemotherapy regimen until death or end of follow-up, whichever is earliest From the index date (first determination of platinum-sensitive recurrence) until death or end of follow-up, whichever is earliest From initiation of each subsequent, post-index therapy line until death or end of follow-up, whichever is earliest

CONTACTS AND LOCATIONS:
Overall Officials: Nicoletta Colombo, MD, Study Director — Steering Committee/Advisory Board Members; Laurence Gladieff, MD, Study Director — Steering Committee/Advisory Board Members; Sven Mahner, MD, Study Director — Steering Committee/Advisory Board Members; Isabel Bover, MD, Study Director — Steering Committee/Advisory Board Members; Jacob Korach, MD, Study Director — Steering Committee/Advisory Board Members
Locations (199):
- Australia (9):
  - Research Site, Ballarat
  - Research Site, Birtinya
  - Research Site, Campbelltown
  - Research Site, East Melbourne
  - Research Site, Mandurah, Western Australia
  - Research Site, South Brisbane
  - Research Site, St Leonards
  - Research Site, Victoria
  - Research Site, Waratah
- Belgium (3):
  - Research Site, Edegem
  - Research Site, Namur
  - Research Site, Sint-Niklaas
- Canada (8):
  - Research Site, Alberta
  - Research Site, Charlottetown
  - Research Site, Mississauga
  - Research Site, Montreal
  - Research Site, Ottawa
  - Research Site, Red Deer
  - Research Site, Toronto
  - Research Site, Vancouver
- France (29):
  - Research Site, Aix-en-Provence
  - Research Site, Ajaccio
  - Research Site, Auxerre
  - Research Site, Besançon
  - Research Site, Béziers
  - Research Site, Bordeaux
  - Research Site, Bourg-en-Bresse
  - Research Site, Brest
  - Research Site, Caen
  - Research Site, Chambéry
  - Research Site, Colombes
  - Research Site, Grenoble
  - Research Site, Libourne
  - Research Site, Longjumeau
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Mont-de-Marsan
  - Research Site, Montbéliard
  - Research Site, Montpellier
  - Research Site, Mulhouse
  - Research Site, Nantes
  - Research Site, Narbonne
  - Research Site, Quimper
  - Research Site, Rennes
  - Research Site, Saint-Pierre-du-Mont
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Villejuif
- Germany (27):
  - Research Site, Bad Godesberg
  - Research Site, Berlin
  - Research Site, Chemnitz
  - Research Site, Cologne
  - Research Site, Düsseldorf
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Frankfurt am Main
  - Research Site, Hagen
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Heilbronn
  - Research Site, Karlsruhe
  - Research Site, Kiel
  - Research Site, Köthen
  - Research Site, Leverkusen
  - Research Site, München
  - Research Site, Nuremberg
  - Research Site, Osnabrück
  - Research Site, Passau
  - Research Site, Ratingen
  - Research Site, Saarlouis
  - Research Site, Stuttgart
  - Research Site, Ulm
  - Research Site, Velbert
  - Research Site, Wetzlar
- Israel (9):
  - Research Site, Afula
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Netanya
  - Research Site, Petah Tikva
  - Research Site, Rehovot
  - Research Site, Saint Holon
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
- Italy (48):
  - Research Site, Alessandria
  - Research Site, Aosta
  - Research Site, Ariano Irpino
  - Research Site, Avellino
  - Research Site, Bari
  - Research Site, Brescia
  - Research Site, Brindisi
  - Research Site, Caltagirone
  - Research Site, Candiolo
  - Research Site, Carbonia
  - Research Site, Castelfranco Veneto
  - Research Site, Castellana Grotte
  - Research Site, Castellaneta
  - Research Site, Catania
  - Research Site, Figline Valdarno
  - Research Site, Franca
  - Research Site, Genova
  - Research Site, Gorizia
  - Research Site, Gravina di Catania
  - Research Site, Ivrea
  - Research Site, Latina
  - Research Site, Latisana
  - Research Site, Lecce
  - Research Site, Lido di Ostia
  - Research Site, Manduria
  - Research Site, Manerbi
  - Research Site, Milan
  - Research Site, Monselice
  - Research Site, Monserrato
  - Research Site, Monza
  - Research Site, Napoli
  - Research Site, Orbassano
  - Research Site, Padua
  - Research Site, Palmanova
  - Research Site, Ponte A Niccheri
  - Research Site, Portogruaro
  - Research Site, Reggio Calabria
  - Research Site, Rieti
  - Research Site, Rionero in Vulture
  - Research Site, Roma
  - Research Site, San Gavino Monreale
  - Research Site, Santorso VI
  - Research Site, Seriate
  - Research Site, Sesto San Giovanni
  - Research Site, Solofra
  - Research Site, Taranto
  - Research Site, Torino
  - Research Site, Trieste
- Netherlands (5):
  - Research Site, Dordrecht
  - Research Site, Enschede
  - Research Site, Leiderdorp
  - Research Site, Nijmegen
  - Research Site, Purmerend
- Portugal (12):
  - Research Site, Barreiro
  - Research Site, Cascais
  - Research Site, Coimbra
  - Research Site, Covilha
  - Research Site, Lisbon
  - Research Site, Martinho Do Bispo
  - Research Site, Portimão
  - Research Site, Porto
  - Research Site, S. Martinho Do Porto
  - Research Site, Santa Maria da Feira
  - Research Site, Setúbal
  - Research Site, Vila Nova de Gaia
- South Korea (2):
  - Research Site, Gyeonggi-do
  - Research Site, Seoul
- Spain (14):
  - Research Site, Alicante
  - Research Site, Alzira, Valencia
  - Research Site, Barcelona
  - Research Site, Elche
  - Research Site, Las Palmas
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Murcia
  - Research Site, Ourense
  - Research Site, Segovia
  - Research Site, Seville
  - Research Site, Terrassa
  - Research Site, Toledo
  - Research Site, Valencia
- Switzerland (14):
  - Research Site, Aarau
  - Research Site, Allschwil
  - Research Site, Baden
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Frauenfeld
  - Research Site, Liestal
  - Research Site, Lucerne
  - Research Site, Rorschach
  - Research Site, Sankt Gallen
  - Research Site, Sion
  - Research Site, Sursee
  - Research Site, Wetzikon
  - Research Site, Zurich
- United Kingdom (19):
  - Research Site, Basingstoke
  - Research Site, Bradford
  - Research Site, Brighton
  - Research Site, Bristol
  - Research Site, Cambridge
  - Research Site, Canterbury
  - Research Site, Glasgow
  - Research Site, Gloucester
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Oxford
  - Research Site, Plymouth
  - Research Site, Reading
  - Research Site, Sheffield
  - Research Site, Southend-on-Sea
  - Research Site, Taunton
  - Research Site, Wales
  - Research Site, Wolverhampton

REFERENCES:
- See also: D0816R00004_CSR_Synopsis_23Feb2017.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2941&filename=D0816R00004_CSR_Synopsis_23Feb2017.pdf